CLINICAL TRIAL: NCT06580223
Title: Aspirin or Rivaroxaban Thromboprophylaxis for Patients With Multiple Myeloma: A Prospective, Multicenter, Open-Label, Randomized Trial
Brief Title: Aspirin or Rivaroxaban Thromboprophylaxis for Patients With Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHCT240465
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Venous Thromboembolism
Keywords: Multiple Myeloma; Venous Thromboembolism; aspirin; rivaroxaban; thromboprophylaxis
MeSH Terms: conditions — Multiple Myeloma; Venous Thromboembolism | interventions — Aspirin; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin,100mg qd, for six months
  Interventions: Drug: Aspirin 100mg
- Rivaroxaban (Experimental): Rivaroxaban, 10mg qd, for six months
  Interventions: Drug: Rivaroxaban 10mg

INTERVENTIONS:
Drug: Aspirin 100mg — Aspirin, enteric coating of tablets, oral administration
  Arms: Aspirin
Drug: Rivaroxaban 10mg — Rivaroxaban, tablets, oral administration.
  Arms: Rivaroxaban

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of aspirin and rivaroxaban in thromboprophylaxis in Chinese MM patients at high risk for MM-associated VTE.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is one of the most common and dangerous complications of Multiple Myeloma (MM). The occurrence of VTE can disrupt treatment plans, compromise patients' quality of life, and even threaten their lives, presenting significant challenges in clinical management. Although several guidelines recommend risk-stratified thromboprophylaxis, there is a deficiency in prospective validation, and most initial studies were conducted in Western cohorts. This prospective, multicenter, open-label, randomized study aims to compare the efficacy and safety of aspirin or rivaroxaban in preventing VTE in Chinese MM patients who are at high risk for VTE.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma (according to Guidelines for the diagnosis and management of multiple myeloma in China (2022 revision))
2. High risk of VTE (according to Expert consensus on the prevention and treatment of multiple myeloma related venous thromboembolism in China (2022))
3. Life expectancy exceeding 12 months
4. Gender: not specified, Age: 18-90 years
5. Serum HIV antigen or antibody negative
6. HCV antibody negative, or HCV antibody positive with HCV RNA negative
7. Echocardiogram shows a left ventricular ejection fraction of ≥50%
8. Ability to sign an informed consent form

Exclusion Criteria:

1. Pregnant women or women who are breastfeeding
2. Active gastrointestinal ulceration
3. Active bleeding
4. When initiating treatment, platelet count below 50 G/L, or with PT prolonged by more than 3 seconds, and APTT prolonged by more than 10 seconds.
5. Abnormal liver function (ALT or AST greater than 3 times the upper limit of normal, or total bilirubin greater than 2 times the upper limit of normal)
6. Abnormal renal function (creatinine clearance < 30 mL/min)
7. Unable to cooperate in completing the clinical trial
8. Already enrolled in other clinical studies
9. Diagnosed with smoldering multiple myeloma or plasma cell leukemia
10. Patients already on antiplatelet therapy for other cardiovascular or cerebrovascular diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of VTE within 6 months | 6 months
  Participants will receive a chest X-ray (or lung CT scan) and a color Doppler ultrasound of the limb blood vessels before the study begins, and then once monthly for the next six months.

SECONDARY OUTCOMES:
Side effects of aspirin and rivaroxaban within 6 months | 6 months
  Testing indicators, including blood routine, urine routine, stool routine, liver and kidney function tests, electrolytes, blood glucose, and blood lipids, will be recorded before the study begins and then once weekly for the next six months. Other observational indicators, such as hemorrhagic events, nausea, vomiting, diarrhea, and abdominal distension, will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided